CLINICAL TRIAL: NCT04859283
Title: Premedication with Intranasal Dexmedetomidine in Sedation of Patients Undergoing Total Knee Arthroplasty
Acronym: TKADEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Teijo Saari, MD, PhD, Professor and Head Physician, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TKADEX
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis; Pain, Postoperative
Keywords: intranasal; dexmedetomidine; multimodal analgesia
MeSH Terms: conditions — Osteoarthritis, Knee; Pain, Postoperative | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX-group (Active Comparator): intranasal dexmedetomidine 1 µg/kg
  Interventions: Drug: Dexmedetomidine
- PLACEBO-group (Placebo Comparator): intranasal saline 10 µL/kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine 1µg/kg will be administered 30min before the induction of anesthesia using a LMA MAD Nasal-device
  Other Names: Dexdor
  Arms: DEX-group
Drug: Placebo — Intranasal saline (10 µL/kg) will be administered 30 min before the induction of anesthesia using a LMA MAD NasalTM -device. The dose is euvolemic to 1 µg/mL dexmedetomidine.
  Other Names: Saline
  Arms: PLACEBO-group

SUMMARY:
This study aims to find out if preoperatively given dexmedetomidine is effective analgesic adjuvant for treating postoperative pain in patients undergoing elective total knee arthroplasty (TKA). Another aim is to determine if premedication with intranasal dexmedetomidine could provide sufficient sedation to alleviate anxiety during TKA.

DETAILED DESCRIPTION:
Patients undergoing total knee arthroplasty (TKA) under spinal anesthesia often request sedation to alleviate anxiety. Dexmedetomidine may be ideally suited to provide sedation during surgery as it offers sedation and analgesia without causing significant respiratory depression. Furthermore, dexmedetomidine has beneficial synergistic interactions with opioids and sedative drugs.

Altogether 80 patients scheduled for elective unilateral TKA under spinal anesthesia will be included in the prospective, randomized and controlled parallel-group study. Patients will be randomized into two groups, forty patients in each group. All patients will receive preoperatively 1000 mg of oral paracetamol as premedication. One group receives a single bolus dose of intranasal 1 ug/kg dexmedetomidine (DEX group) and the other group receives euvolemic dose (10 µL/kg) of saline (PLACEBO-group).

Spinal anesthesia will be performed using bupivacaine (5 mg/mL) using 2.0-2.5 mL dose, the amount depending on the clinical judgement of the anesthesiologist responsible for the patient. If patient needs additional analgesic after spinal anesthesia, 50 µg dose of intravenous fentanyl or 3-5 mg of intravenous midazolam may be administered intraoperatively.

Postoperative pain management in the surgical ward includes oral paracetamol 1000 mg every 8 hours, and from the first postoperative day onwards patients receive oral naproxen/esomeprazole 500/20 mg twice a day. Oral oxycodone (5-10 mg) will be used, if the pain (measured with numerical rating scale, NRS, min 0, max 100, higher scores mean worse outcome) is moderate or intense (NRS>30) after paracetamol and naproxen.

Postoperative pain (NRS) and opioid consumption (mg) will be measured and analysed together with intraoperative sedative used (mg, midazolam and/or fentanyl allowed).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is scheduled for elective unilateral total knee arthroplasty (TKA) under spinal anesthesia
2. Fluent skills in finnish language (to understand the given information and to be able to give informed consent and communicate with the study personnel)
3. Age between 35 and 80 years
4. Weight between 50 and 100 kg
5. American Society of Anesthesiologists status 1-3
6. Written informed consent from the patient

Exclusion Criteria:

1. A previous history of intolerance to the study drug or related compounds and additives
2. Disease or condition affecting patient's ability to give written informed consent
3. Existing or recent disease possible affecting absorption, distribution, metabolism, excretion or response to the study drug
4. History of severe cardiac disease (valvular insufficiency, severe left ventricular dysfunction) or abnormal ECG rhythm (bradycardia < 50/min, 2nd or 3rd degree atrioventricular-block, pacemaker)
5. Preoperative systolic blood pressure <110 mmHg
6. Chronic use of strong opioids, pregabalin, gabapentin, amitriptyline or duloxetine
7. Participation in any other study concomitantly or within one month prior to the entry into this study
8. Clinically significant abnormal findings in physical examination or laboratory screening
9. Pregnancy or breastfeeding
10. Use of any drugs known to cause enzyme induction or inhibition for a period of 30 days prior to the study, use of any natural products (including grapefruit products) for at least 14 days prior to the study and caffeine containing products for at least 24 hours prior to the study. The use of regular doses of paracetamol is allowed.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in numerical rating scale (NRS 0-100 mm, min 0, max 100, higher score means worse outcome) | 24 hours
  Number of patients with visual rating scale value under 30 mm
Change in intraoperative sedatives (mg) administered | From anesthesia induction to the end of surgery.
  Change from baseline midazolam and fentanyl consumption (mg)
Change in opioid consumption (mg) postoperatively | 24 hours
  Change from baseline opioid consumption (mg) postoperatively at 24 hours

SECONDARY OUTCOMES:
Change (mmHg) in hemodynamic parameter (blood pressure) | 24 hours
  More than 30% change from the baseline in the blood pressure (measured in mmHg)
Change (%) in respiratory parameter (peripheral oxygen saturation, SpO2) | 24 hours
  More than 10% change from the baseline in the SpO2 (measured %)
Number of patients with adverse events as a measure of safety and tolerability | 24 hours
  Number of patients with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Suvi-Maria Tiainen, MD, Principal Investigator — Turku University Hospital, University of Turku
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital and University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiainen SM, Heinonen H, Koskinen A, Makela S, Laitio R, Loyttyniemi E, Makela K, Saari TI, Uusalo P. Premedication with intranasal dexmedetomidine in patients undergoing total knee arthroplasty under spinal anaesthesia (TKADEX)-a prospective, double-blinded, randomised controlled trial. BJA Open. 2025 Mar 3;13:100382. doi: 10.1016/j.bjao.2025.100382. eCollection 2025 Mar. PMID 40114985